CLINICAL TRIAL: NCT02966821
Title: A Phase II, Single-arm, Open-label, Multicenter Study to Assess the Efficacy and Safety of Surufatinib as a Second-line Treatment in Patients With Surgically Unresectable or Metastatic Biliary Tract Carcinoma
Brief Title: Study of Surufatinib as Second-line Treatment in Patients With Biliary Tract Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-012-00CH1
Record Dates: First submitted 2016-11-11; First posted 2016-11-17 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Biliary Tract Cancer
Keywords: Surufatinib; Biliary Tract Cancer; Second-line
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surufatinib (Experimental): Surufatinib 300mg once-daily
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Patients receive oral Surufatinib at a dose of 300mg/d within 1 hour after breakfast (once-daily dosing continuously, every 28-day treatment cycle)
  Other Names: HMPL-012 and Sulfatinib

SUMMARY:
A phase II, single-arm, open-label, multicenter study to assess the efficacy and safety of Surufatinib as a second-line treatment in patients with surgically unresectable or metastatic biliary tract carcinoma

DETAILED DESCRIPTION:
This study adopt Simon's two-stage designs method based on the primary endpoint of 16-week PFS rates. In the first stage, 16 patients will be recruited. If there are 3 or fewer patients without progression or death out of these 16 patients at week 16, the study will be stopped. Otherwise, 16 additional patients will be accrued for a total of 32 evaluable patients.

Surufatinib will be orally administered within 1 hour after breakfast once a day (QD) for every 28-day treatment cycle until disease progression, death, intolerable toxicity or other protocol specified end-of-treatment criteria is met (which comes first).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written Informed Consent Form (ICF) prior to any study specific procedures
2. Aged at least 18 years
3. Histologically or cytologically confirmed advanced BTC that was surgically unresectable or metastatic, including extrahepatic cholangiocarcinoma (EHCC), intrahepatic cholangiocarcinoma (IHCC) or gallbladder biliary carcinoma (GBC)
4. First-line prior treatment of cytotoxic chemotherapy, treatment failure or intolerable toxicities
5. ECOG 0-1
6. Patients must have measurable lesions

Exclusion Criteria:

1. Anti-tumor therapy received within 4 weeks prior to initiation of study treatment
2. Previous therapy with approved or investigational anti-VEGF (or VEGFR) tyrosine kinase inhibitors or monoclonal antibody
3. Liver metastases ≥50% of liver volume
4. Child-Pugh classification score of liver function> 7
5. History or presence of a serious hemorrhage (>30 ml within 3 months), hemoptysis (>5 ml blood within 4 weeks) or a thromboembolic event (including transient ischemic attack and/or stroke events) within 12 months
6. Active malignancy (except for definitively treated basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 5 years
7. Patients receive CYP3A4 potent inducer or inhibitors within 2 weeks
8. Pregnancy ( positive pregnancy test before the first dose of study treatment) or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at Week 16 | Progression-free survival (PFS) rate at Week 16
  Proportion of patients without PD or death at Week 16

SECONDARY OUTCOMES:
Adverse events evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 | From first dose to within 30 days after the last dose
  AE monitored from the first dose to within 30 days after the last dose
Clinically significant laboratory, vital sign or physical examination abnormalities, electrocardiogram (ECG) and echocardiogram changes | From first dose to within 30 days after the last dose
  Safety parameters monitored from the first dose to within 30 days after the last dose
Objective response rate (ORR) | 6 months after the last patient enrolled
  Proportion of patients with a best overall CR and PR per RECIST v1.1
Disease control rate (DCR) | 6 months after the last patient enrolled
  Proportion of patients whose best overall response from baseline is either a CR, PR or SD per RECIST v1.1
Duration of response (DoR) | 6 months after the last patient enrolled
  The time from the first time that the objective response reaches CR or PR, whichever comes first, until the occurrence of PD or death
Progression-free survival (PFS) | 6 months after the last patient enrolled
  The time from the start date of study drug until the date of objective disease progression or death
Overall survival (OS) | 6 months after the last patient enrolled
  The time interval between the start date of study drug and the date of death (any cause)

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, Prof., Principal Investigator — The 307th Hospital of Military Chinese People's Liberation Army
Locations (5):
- China (5):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The 307th Hospital of Military Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Heilongjiang Cancer Hospital, Harbin, Heilongjiang
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Tianjin medical university cancer institute&hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No